CLINICAL TRIAL: NCT04101838
Title: B Cell and Antibody Response to Seasonal Influenza Vaccines in Younger and Older Adults
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, James Kobie, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-300003914
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Influenza
Keywords: vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Fluzone High-Dose; fluad vaccine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be blinded to which vaccine they receive until immediately after vaccination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Fluzone Younger (Active Comparator): 10 adults 18-50 years old, will receive a single dose of the Fluzone influenza vaccine each year for two sequential years
  Interventions: Drug: Fluzone
- Flucelvax (Active Comparator): 10 adults 18-50 years old, will receive a single dose of the Flucelvax influenza vaccine each year for two sequential years
  Interventions: Drug: Flucelvax
- Fluzone Older (Active Comparator): 10 adults 65-80 years old, will receive a single dose of the Fluzone influenza vaccine
  Interventions: Drug: Fluzone
- Fluzone High Dose (Active Comparator): 10 adults 65-80 years old, will receive a single dose of the Fluzone High-Dose influenza vaccine
  Interventions: Drug: Fluzone High-Dose
- Fluad (Active Comparator): 10 adults 65-80 years old, will receive a single dose of the Fluad influenza vaccine
  Interventions: Drug: Fluad

INTERVENTIONS:
Drug: Fluzone — inactivated seasonal influenza vaccine
  Other Names: influenza vaccine
  Arms: Fluzone Older; Fluzone Younger
Drug: Flucelvax — inactivated seasonal influenza vaccine
  Other Names: influenza vaccine
  Arms: Flucelvax
Drug: Fluzone High-Dose — inactivated seasonal influenza vaccine
  Other Names: high dose influenza vaccine
  Arms: Fluzone High Dose
Drug: Fluad — inactivated seasonal influenza vaccine
  Other Names: adjuvanted influenza vaccine
  Arms: Fluad

SUMMARY:
This study will examine how various FDA-approved seasonal influenza vaccine types, used in a manner consistent with their approved use, impact the characteristics of influenza specific antibodies in humans, and how these responses differ based on age and prior immunization history.

DETAILED DESCRIPTION:
This study is particularly focused on studying antibodies, a protein in blood that react with foreign substances (such as bacteria and viruses) to help eliminate them. This study will examine antibodies and the cells that they are produced by, B cells that develop in response to the influenza vaccine.

The majority of antibodies that develop following seasonal influenza vaccine are highly specific for particular influenza strain that comprises the influenza vaccine, necessitating the annual reformulation of the influenza vaccine to match strains expected to be in circulation for the upcoming season. This is problematic, and strategies to develop an influenza vaccine that can promote the robust and persistent development of antibodies that are effective against a wide range of influenza strains are needed. One potential strategy is to promote antibody responses targeting the neuraminidase (NA) protein of influenza. NA is more highly conserved across influenza viruses as compared to the hemagglutinin (HA) protein which is the major component of the influenza vaccine. Thus understanding how differences in seasonal influenza vaccines may influence the quality and breadth of HA and NA specific antibodies is of importance in the development of more effective influenza vaccines.

There are several FDA-approved seasonal inactivated influenza vaccines (IIVs) and it remains unknown the extent to which they may induce HA and NA-specific B cells and antibodies, and particularly those that may have broad protective activity against influenza. Differences in the various seasonal IIVs, such as how they were produced, their dose, and the immune stimulating components (adjuvant) they contain may influence the HA and NA-specific response. The two major types of seasonal IIV approved for adults are IIV that is comprised of inactivated influenza virus that was grown in chicken eggs (e.g. Sanofi Fluzone, IIV), and the other comprised of inactivated influenza virus that was grown in cell culture (e.g. Seqirus Flucelvax, cc-IIV). Additionally, for adults 65 years and older, High Dose Fluzone (HD-IIV3), and Sequris Fluad IIV, which includes an adjuvant (a-IIV3). This study will evaluate the relative induction of HA and NA-specific antibodies and B cells from adults immunized with these various seasonal influenza vaccines, and how these responses may change after each year, and differ in older adults who may have a different past exposure history to influenza compared to younger adults. The seasonal influenza vaccines will be given as standard of care, in populations they are approved for, and administered in approved dose and route.

ELIGIBILITY:
Inclusion Criteria:

* Participation in ancillary clinical research study
* Able to give informed consent
* Age 18-50 years old for Arm 1 and Arm 2
* Age 65-80 years old for Arm 3, Arm 4, and Arm 5
* Weight of at least 110 lbs as determined by self-reporting

Exclusion Criteria:

* Inability to give informed consent
* Refusal or inability to have blood drawn or participate in study procedures
* Previous adverse reaction to influenza vaccine or medical history contraindicated for receiving influenza vaccine, including but not limited to:

  1. History of Guillain-Barre Syndrome
  2. History of egg allergy
  3. History of gelatin allergy
  4. History of moderate to severe illness with or without fever within 6 weeks of receipt of influenza vaccine
* Previous receipt of influenza vaccine outside of study within current season
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Participant has any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgement of the investigator would interfere with, or serve as a contraindication to the planned procedure(s).
* These following criteria are used for scientific reasons, and not safety reasons. Specifically, the criteria are used to obtain a population that is healthy and less likely to have conditions that may influence the immune system:

  1. No recent respiratory infections in the past 4 weeks at time of vaccination
  2. Malignancy
  3. Evidence of Inflammation: Systemic Lupus Erythematosis, Rheumatoid Arthritis, Polymyositis, Dermatomyositis, Scleroderma, Crohn's Disease, Ulcerative Colitis.
  4. Lymphoproliferative Disorder
  5. Known Immunodeficiency
  6. Myocardial Infarction <6 months
  7. Cerebral Vascular Accident
  8. Peripheral Vascular Disease- recannulation <6months
  9. Cardiac Insufficiency - congestive heart failure
  10. Hypertension with increased blood urea nitrogen (BUN)
  11. Renal Failure
  12. Dementia
  13. Alcoholism (defined as >17 drinks/week)
  14. Drug Abuse (excluding marijuana)
  15. HIV positive
  16. History of hepatitis
  17. History of immunization within 4 weeks of study participation or plan to receive non- IIV vaccination within 4 weeks of receiving IIV
  18. Moderate to severe illness at time of enrollment
* Donations of blood in the 8 weeks prior to enrollment which, combined with expected volumes to be drawn for this study, would exceed 450 mL in an 8 week period.
* Current pregnancy at time of enrollment or pregnancy within last 4 months
* Active or planned breastfeeding during study participation
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Hemagglutinin antibody | 3 months after vaccination
  hemagglutinin plasma antibody titer
Neuraminidase antibody | 3 months after vaccination
  Neuraminidase plasma antibody titer

SECONDARY OUTCOMES:
Hemagglutinin Memory B cell ELISPOT Response | 3 months after vaccination
  hemagglutinin-specific memory B cells
Neuraminidase Memory B cell ELISPOT Response | 3 months after vaccination
  Neuraminidase-specific memory B cells

CONTACTS AND LOCATIONS:
Overall Officials: James J Kobie, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No